CLINICAL TRIAL: NCT03466437
Title: Survival of Abutment Teeth of Removable Partial Dentures Rehabilitated With Post-retained Restorations: Randomized Clinical Trial
Brief Title: Post-retained Restorations for RPD Abutments
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Pelotas (Other)
Responsible Party: Principal Investigator, Maximiliano Sergio Cenci, Professor, Federal University of Pelotas
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PPGO021
Record Dates: First submitted 2018-02-28; First posted 2018-03-15 (Actual); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Tooth, Nonvital; Composite Resins; Metal Ceramic Restorations; Denture, Partial, Removable; Post and Core Technique
MeSH Terms: conditions — Tooth, Nonvital

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Glass-fiber post + composite resin restoration (Experimental)
  Interventions: Device: Glass-fiber post and composite resin restoration
- Glass-fiber post + metalceramic crown (Experimental)
  Interventions: Device: Glass-fiber post and metalceramic crown
- Cast-metal post + metalceramic crown (Active Comparator)
  Interventions: Device: Cast-metal post and metalceramic crown

INTERVENTIONS:
Device: Glass-fiber post and composite resin restoration — Patients will receive a glass-fiber and composite resin restoration followed by removable partial denture fabrication
  Arms: Glass-fiber post + composite resin restoration
Device: Glass-fiber post and metalceramic crown — Patients will receive a glass-fiber and metalceramic crown followed by removable partial denture fabrication
  Arms: Glass-fiber post + metalceramic crown
Device: Cast-metal post and metalceramic crown — Patients will receive a cast-metal post and metalceramic crown followed by removable partial denture fabrication
  Arms: Cast-metal post + metalceramic crown

SUMMARY:
This study will be a controlled, randomized, parallel group trial where the survival rate of direct and indirect restorations on removable partial denture abutment teeth will be assessed. For this, individuals with widely destroyed teeth and need for endodontic treatment, with at least one remaining dentin wall, adjacent to edentulous spaces in Kennedy Classes I and II will be selected. After the minimum period of one year the teeth will be reassessed through clinical and radiographic examination annually.

All patients will receive oral hygiene instructions, caries disease control and endodontic treatment according to the need of each case. Prior to post cementation, patients will receive endodontic treatment through routine techniques that include use of rubber dam, mechanized instrumentation with NaOCl 2%, gutta percha and endodontic cement filling and condensation by the McSpadden technique. The preparation for post space will be done with a specific bur compatible with the diameter of root canal, and the same preparation cast post and cores. The glass-fiber posts (will be cleaned with 70% alcohol and receive silane application.

The clinical protocol for direct restoration and confection of the composite resin core will occur in the same way, using the same materials: the dental structure will be etched with 37% phosphoric acid and rinsed, followed by the adhesive system and fabrication of the restoration by incremental technique according to the manufacturer's recommendations. It is important to emphasize that the direct restorative procedure will be carried out in the same consultation of the glass-fiber post cementation.

In order to make the cast metal cores, the indirect impression technique will be done with prefabricated pins associated with addition silicone. In this technique, the lightweight material will be inserted into root canal and then, the pin will be introduced into the canal. Next, a prefabricated tray with the heavy and light material will be positioned for removal of the assembly, being removed after the setting time determined by the manufacturer. The mold obtained will be sent to the dental technician for cast post and core fabrication. All posts will be cemented under rubber-dam isolation using self-adhesive resin cement.

In teeth where randomization is a metalceramic crown, first the composite resin or metal core will be prepared with a 3216 drill, in order to obtain 1.5mm wear on the proximal and free faces and 2mm on the occlusal surface. The margin design in form of a chamfer, preferably at the gingival level whenever possible. The impression procedure will be carried out using a molding cap and polyether, which will be removed in a tray with irreversible hydrocolloid. A temporary crown will also be made for the patient. The metallic infrastructure will be tested in order to verify its adaptation and transferred in irreversible hydrocolloid molding for later ceramic application. After application of the ceramic, the laying and adaptation of the prosthetic piece will be conferred, being the crown luted with self-adhesive resin cement.

Once the restoration / crown of the abutment tooth has been made, the treatment will continue with the preparation of the removable partial denture. The teeth will always be prepared in the mesial proximal area. The delivery of the removable partial denture will be considered the baseline of the study. At this moment, the necessary adjustments and subsequent control of the prosthesis will be made after 24, 72 hours, a week and 15 days in order to check for possible flaws. After 6 months and 1 year of delivery of the removable partial denture, all patients will be recalled for clinical and radiographic evaluation of prostheses / restorations and oral hygiene conditions. This monitoring will be conducted by two evaluators until the end of the trial.

All clinical procedures will follow pre-established protocols and the data of each patient and intervention will be recorded in the individual patient file.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with good general and oral health;
* unilateral or bilateral free-end edentulism (Kennedy Classes I and II), which have adjacent abutments to edentulous space requiring endodontic treatment and at least 1 (one) remaining dentin wall and requiring intraradicular retention, with adequate bone support;
* minimum 18 years old;
* Knife-tipped alveolar ridges may be included in the study after trimming if the abovementioned criteria are met.

Exclusion Criteria:

* Untreated periodontal disease;
* poor oral hygiene;
* periapical lesion that does not respond to conventional endodontic treatment;
* abutment teeth with mobility greater than grade I;
* lack of prosthetic space due to extrusion of the opposing teeth;
* allergy to the materials used in the removable partial denture;
* absence of occlusal contacts in the antagonist arch;
* patients who are participating in other clinical trials;
* patients who have complete denture opposing the site;
* financial restrictions;
* unable to be followed for a minimum period of 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2018-02-28 (Actual); Primary Completion 2019-02 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Direct Abutment Tooth Survival | Changes from baseline to 3 years of clinical function
  Main outcome will be assessed considering loss (extraction) or maintenance of each restored tooth.
  In order to simplify outcome measure, data for this outcome will be represented as "Tooth loss" (Yes or No)
Crown dislodgment | Changes from baseline to 3 years of clinical function
  In any case that metalceramic crown moves from cemented position, this outcome will be assessed as: "Presence of Crown Dislodgment" (Yes or No)
Post debonding | Changes from baseline to 3 years of clinical function
  In any case that post (glass-fiber or cast-metal post) debond from root canal, this outcome will be assessed as: "Presence of Post Debonding" (Yes or No)
Restoration Fracture | Changes from baseline to 3 years of clinical function
  Described as any fracture of restorative material, this outcome will be assessed as: "Presence of Restoration Fracture" (Yes or No)
Post and core fracture | Changes from baseline to 3 years of clinical function
  Clinical assessment of restored teeth will present data from this outcome as: "Presence of Post and Core Fracture" (Yes or No)
Root fracture | Changes from baseline to 3 years of clinical function
  Clinical assessment of restored teeth will present data from this outcome as: "Presence of Root Fracture" (Yes or No)
Secondary caries | Changes from baseline to 3 years of clinical function
  Clinical assessment of restored teeth will present data from this outcome as: "Presence of secondary caries" (Yes or No)

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Pelotas - School of Dentistry, Pelotas, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No